CLINICAL TRIAL: NCT06278025
Title: Comparison of Deep Cervical Flexor Muscle Strength and Endurance in Patients With and Without Neurogenic Dysphagia
Brief Title: Dysphagia and Deep Cervical Flexor Muscles
Status: Completed | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: GO 19/833
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia; Neurological Disorder
MeSH Terms: conditions — Deglutition Disorders; Nervous System Diseases | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with dysphagia (study): In the modified barium swallowing study, liquid in the amount of 5 ml was used because it is the optimal amount to monitor physiological events during swallowing . The Penetration Aspiration Scale (PAS) was used to determine the dysphagia severity. The PAS is an 8-point scale describing the degree and nature of laryngeal penetration and aspiration, where a score of 1 refer to 'No penetration or aspiration- No entry of material into the airway', and 8 refer to 'Airway aspiration- Material enters the trachea with no attempt to clear'. According to the MBSS, patients who received a PAS score of 1 were included in the group without dysphagia (control group), and those received a PAS score between 2 and 8 were included in the group with dysphagia (study group).
  Interventions: Diagnostic Test: assessment
- patients without dysphagia (control): In the modified barium swallowing study, liquid in the amount of 5 ml was used because it is the optimal amount to monitor physiological events during swallowing . The Penetration Aspiration Scale (PAS) was used to determine the dysphagia severity. The PAS is an 8-point scale describing the degree and nature of laryngeal penetration and aspiration, where a score of 1 refer to 'No penetration or aspiration- No entry of material into the airway', and 8 refer to 'Airway aspiration- Material enters the trachea with no attempt to clear'. According to the MBSS, patients who received a PAS score of 1 were included in the group without dysphagia (control group), and those received a PAS score between 2 and 8 were included in the group with dysphagia (study group).
  Interventions: Diagnostic Test: assessment

INTERVENTIONS:
Diagnostic Test: assessment — DCF Muscle Strength Evaluation
  DCF muscle strength was determined using the 5-step Craniocervical Flexion Test (CCFT) performed with a Chattanooga Stabilizer ™ Pressure Biofeedback Unit which was developed by Jull et al. [33, 34]. The CCFT is based on the craniocervical flexion movement, which is provided by DCF muscle contraction. The CCFT includes 5 pressure increments starting with 20mmHg.Activation score ranges from 0 to 10. The performance index is determined by both the highest pressure level and the number of repetitions.
  Evaluation of the DCF Endurance The DCF endurance test, which is a valid and reliable method, was used to measure DCF muscle endurance [36]. Conducted in supine, endurance is measured by calculating the time (in seconds) an individual can raise their head at minimal flexion angle.

SUMMARY:
Cervical posture is vital for normal swallowing function. Changes in cervical posture during swallowing alter the bolus flow and swallowing kinematics through changes in gravity and oropharyngeal space. The hyoid bone does not articulate with any bone, so it requires adequate tension of the hyolaryngeal complex and proper cervical postural alignment to maintain its stabilization and position. Changes in cervical posture and stabilization can cause changes in hyoid bone position and kinematics through muscles and ligaments which may lead to decrease in hyoid elevation, loss of optimal strength of the suprahyoid and infrahyoid muscles due to disrupted length-tension relationship, and an increased risk of aspiration due to insufficient laryngeal elevation. Further, deterioration in cervical posture and decreased stabilization resulting from cervical muscle weakness or/both endurance could affect the control and strength of masticatory muscles, tongue muscles and suprahyoid - infrahyoid muscles, which are involved in swallowing function. Whereby DCF weakness gives rise to inadequate cervical stabilization, change in hyoid bone stabilization, alterations in suprahyoid and infrahyoid muscle function, and decreased laryngeal elevation may adversely affect the normal function of the swallowing related muscles. Thus, decreased cervical stabilization, which is often seen in neurological diseases, may be related to neurogenic dysphagia. Given the known changes in cervical stabilization as a consequence of neurologic injury, the additional impact on swallowing or a potentially already neurologically-disordered swallow is considered. Thus, loss of cervical stabilization may be one of the factors affecting dysphagia in patients with neurological diseases providing more information on all potential factors contributing to swallow impairment, potentially leading to more targeted and effective swallowing interventions. However, there is no study investigating the role of the DCF muscles in dysphagia. Therefore, the aim of the present study was to comparison of deep cervical flexor muscle strength and endurance in patients with and without neurogenic dysphagia.

ELIGIBILITY:
Inclusion Criteria:

- diagnosis of neurological disease, age range inclusive of 18-65 years , independent sit-to-stand, prior consultation for dysphagia, and underwent a Modified Barium Swallowing Study (MBSS).

Exclusion Criteria:

* neck pain complaints in the previous 30 days history of cervical surgery and head and neck cancer, cervical pathology involving the neck region such as cervical disc herniation or radiculopathy presence of cervical osteophytes and/or cervical kyphosis detected in the MBSS, history of rheumatic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants aged between 18 - 65 and diagnoses neurological disease will included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
dcf muscle strenght | 1 day
dcf endurance | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: sena N begen, Study Chair — Atilim University, Faculty of Health Sciences Department of Physiotherapy and Rehabilitation; selen serel arslan, Study Director — Hacettepe University Faculty of Physical Therapy and Rehabilitation Ankara, TURKEY
Locations (1):
- Atilim University, Ankara, Incek, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided